CLINICAL TRIAL: NCT02881112
Title: An Open-Label, Non-Controlled Study to Evaluate Outcomes of Pulsed Electromagnetic Field (PEMF) Therapy in Subjects With Various Pain Etiologies
Brief Title: A Registry Study to Evaluate Outcomes of PEMF Therapy in Subjects With Various Pain Etiologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBI.2015.005
Record Dates: First submitted 2016-06-30; First posted 2016-08-26 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Treatment Arm (Experimental): Treatment with Provant Therapy System
  Interventions: Device: Provant Therapy System

INTERVENTIONS:
Device: Provant Therapy System — Treatment with the Provant Therapy System

SUMMARY:
The study is an open-label, non-controlled study of the safety and effectiveness of investigator determined Provant therapy in subjects with pain and/or edema from various pain etiologies. Information collected in the study will be entered into a registry database.

DETAILED DESCRIPTION:
This is an open-label, non-controlled trial in subjects with various pain etiologies at multiple centers in the US. Eligible subjects will include those ≥ 22 years of age that have been deemed appropriate for treatment with Provant by the study investigator (prescriber). Subjects will treat based on the treatment prescribed (location, frequency, duration) by the study investigator.

Data from assessments administered as part of standard of practice will be obtained at baseline and, at a minimum, at the end of treatment. If the investigator administers additional assessments during the course of treatment, the data will be collected.

Safety will be assessed during office visits and through review of AE reports and concomitant treatments and medications. All concomitant drug or non-drug treatments used during the study will be recorded.

Information collected in the study will be entered into a registry database.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is greater than or equal to 22 years.
2. Subject has pain (chronic or acute) and/or edema that the prescriber deems treatment with Provant is warranted.
3. Subject is willing and able to give written informed consent.
4. Female subjects must be post-menopausal, surgically sterile, abstinent, or practicing (or agree to practice) an effective method of birth control if they are sexually active for the duration of the study. (Effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier methods, and/or male partner sterilization).

Exclusion Criteria:

1. Subject requires or anticipates the need for surgery of any type during the duration of treatment.
2. Subject has received any investigational drug or device within 30 days or 5 half-lives of the drug, whichever is longer, prior to the Screening Visit or is enrolled in another clinical trial.
3. Subject has used systemic corticosteroids within 2 months of the Screening Visit.
4. Subject has a history of a solid tumor that is not in complete remission for greater than 2 years other than successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin in the treatment area.
5. Subject has a history of blood cancer (e.g., leukemia, lymphoma, multiple myeloma).
6. Subject has a serious psychosocial co-morbidity.
7. Subject has a history of drug or alcohol abuse within one year prior to the Screening Visit.
8. Subject has an implanted pacemaker, defibrillator, neurostimulator, spinal cord stimulator, bone stimulator, cochlear implant, or other implanted device with an implanted metal lead(s).
9. Subject is currently pregnant or planning on becoming pregnant during the treatment period.
10. Subject has been previously treated with the Provant Therapy System.
11. Subject is unwilling or unable to follow study instructions, or comply with the treatment regimen and study visits.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - AOC-Research, LLC, Birmingham, Alabama
  - Coolbody Contours, Scottsdale, Arizona
  - Scottsdale Center for Women's Health, Scottsdale, Arizona
  - Coastal Orthopedics & Sports Medicine, Bradenton, Florida
  - Injury Care Research, LLC, Boise, Idaho
  - Exodus Pain Clinic, Meridian, Idaho
  - Biogenesis Group, LLC, Ypsilanti, Michigan
  - Spokane Joint Replacement Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment Arm
Started | 180
Completed | 152
Not Completed | 28

BASELINE CHARACTERISTICS:
Arm/Group | Active Treatment Arm
Number analyzed (Participants) | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 105
  >=65 years | 75
Age, Continuous [Mean (Full Range); unit: Years] | 60.48 [24 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124
  Male | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 153
  Unknown or Not Reported | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 149
  More than one race | 1
  Unknown or Not Reported | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 180

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Assessment
Description: Change in Pain from Baseline/Pre-treatment to End of Treatment/Last Available Observation. Pain captured using NPRS, 0-10 scale were 0 = no pain and 10 = worst pain, given to subjects as part of a daily diary.
Time Frame: Pain scores collected daily, up to 20 weeks.
Population: Subjects recording both a Baseline and End of Study score were included in the NPRS analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment Arm
Number analyzed (Participants) | 75
score on a scale | -2.785 (3.3039)

ADVERSE EVENTS:
Time Frame: Through end of treatment, up to 20 weeks.
Arm/Group | Active Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/180
Serious Adverse Events (participants affected / at risk) | 0/180
Other Adverse Events (participants affected / at risk) | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication Rights. Independent analysis and/or publication of data generated or arising from the performance of this Agreement is not permitted without the prior written consent of Regenesis. Such consent may be contingent on Regenesis' review and approval of any proposed analysis and manuscript. Institution will retain the right to review and analyze the database created from this study for its own scientific purposes so long as such scientific purposes are non-commercial in nature.

DOCUMENTS (2):
  • Study Protocol: Study Protocol (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT02881112/Prot_002.pdf
  • Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT02881112/SAP_003.pdf